CLINICAL TRIAL: NCT00530582
Title: Progesterone Reduces Wakefulness in Sleep EEG and Has no Effect on Cognition in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Collaborators: Dr. Kade/Besins Pharma GmbH, Rigistr. 2, 12277 Berlin (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KAD 108 ex
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Healthy; Postmenopausal
Keywords: progesterone, postmenopause, sleep-EEG
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: progesterone — 300mg progesterone /placebo each for 21 days
  Other Names: Utrogest/ Utrogest Placebo Ch.-B.: 0503

SUMMARY:
Sleep is impaired in postmenopausal women (difficulty falling asleep, frequent awakenings). Progesterone prompted benzodiazepine-like effects on sleep EEG in young normal male subjects.

Aim of this study was to test if replacement therapy with progesterone improves sleep after menopause.

Design, Setting, and Participants: A double blind cross-over design study with 2 treatment intervals of 21 days duration separated by a 2 weeks washout was performed. A oral dose of 300mg micronized progesterone was given each for 21 days. At the beginning and the end of the two intervals a sleep EEG was recorded and cognitive performance was assessed in 10 healthy postmenopausal women (age: 54-70 yrs).

DETAILED DESCRIPTION:
Objectives/ Mode of administration: To characterise the effects of progesterone in a dose of 300mg each for 21 days on changes of sleep EEG and cognition in postmenopausal healthy women, in comparison with placebo.

Methodology:The study was performed as double blind randomized placebo controlled crossover design with two treatment intervals of 21 days duration separated by 2 weeks washout. Progesterone was administered as tablets in a dose of 300mg each for 21 days. At the beginning and the end of the two intervals a sleep EEG was recorded after one night of adaptation to laboratory conditions, during which EEG electrodes were attached without recording an EEG.For the registration nights the subjects arrived at the sleep laboratory at 21.00 h. Sleep EEG was recorded from 23.00 h until 07.00 h hours next morning.Cognitive performance was tested after the registration nights at 09.00h.All pharmacodynamic investigations were carried out in the sleep laboratory of the Max Planck Institute of Psychiatry in Munich.

Main criteria for inclusion: Subjects consisted of 10 healthy women (age: range 54-70 years) who entered the study after passing rigid psychiatric, physical and laboratory examinations. They had been drug free at least 4 weeks. Reasons for exclusion from the study were: psychiatric disorder in the subjects own or family history, including dementia or other cognitive impairment; recent stressful life events; substance abuse; a transmeridian flight during the last three months; shift work; medical illness; and aberrations in blood chemistry or in the waking EEG or electrocardiogram.All subjects underwent a polysomnographic examination in the sleep laboratory before entering the study to exclude sleep disorder including sleep related respiratory disorders and sleep related movement disorders.

Statistical methode: Expolatory and inferential statistical analysis of certain aggregated sleep variables after classifying the sleep EEG in dinstinct stages according to Rechtschafen/Kales and of the results of EEG spectral analysis. Inferential statistics were based on multivariate analyses of variance (MANOVAs) with treatment as influential factor and on one sample t-tests for placebo related power changes of progesterone in non-REM sleep as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female elderly subjects
* Age between 55-70 years
* Normal physical examination including a neurological and gynecological examination
* Medical history without major or chronic diseases (e.g. diabetes, heart failure, hepatitis)
* No previous psychiatric or chronic neurological disorder (e.g. schizophrenia, epilepsy)
* Normal standard electrocardiograpy (ECG)
* Normal laboratory results
* Body Mass Index <30
* Normal sleep EEG concerning restless leg and sleep apnoe syndrom
* Normal EEG, according to the guidelines of the Deutsche EEG Gesellschaft (German EEG Society)
* Written informed consent
* Written consent from the gynecologist, who examined the subjects, that there is no contradiction for the oral application of Utrogest

Exclusion Criteria:

* Gastrointestinal disorder
* Gynecological disorder
* Heart and lung disorder
* Liver and kidney disorders
* Creatinin serum >2,5 mg%
* Thyroid diseases
* Psychiatric disorders
* Psychiatric disorder in the family history
* Peripheral and central nervous system disorder
* Metabolic diseases
* Endocrine diseases
* Muscular or dermatological diseases
* Haematological diseases
* Smoker

Further exclusion criteria were:

* Sleeping disorder
* Shift work
* Transmerdian flight in the last three months
* Malignant diseases
* Acute infective diseases
* Clinically relevant allergies
* Lack of compliance to study procedures
* Participation in another clinical study within the last 4 month

Ages: 54 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-11; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
sleep-EEG parameters

CONTACTS AND LOCATIONS:
Overall Officials: Axel Steiger, Prof., MD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany

REFERENCES:
- [Background] Dzaja A, Arber S, Hislop J, Kerkhofs M, Kopp C, Pollmacher T, Polo-Kantola P, Skene DJ, Stenuit P, Tobler I, Porkka-Heiskanen T. Women's sleep in health and disease. J Psychiatr Res. 2005 Jan;39(1):55-76. Ehlers CL, Kupfer DJ. Slow-wave sleep: do young adult men and women age differently? J Sleep Res. 1997 Sep;6(3):211-5. Friess E, Tagaya H, Trachsel L, Holsboer F, Rupprecht R. Progesterone-induced changes in sleep in male subjects. American Journal of Physiology: Endocrinology & Metabolism 1997; 272:E885-E891. Grön G, Friess E, Herpers M, Rupprecht R. Assessment of cognitive performance after progesterone administration in healthy male volunteers. Biol Psychiatry 1997; 35:147-151. Heuser G, Ling GM, Kluver M. Sleep induction by progesterone in the pre-optic area in cats. Electroencephalography & Clinical Neurophysiology 1966; 22:122-127. Lancel M, Faulhaber J, Schiffelholz T, Romeo E, Di Michele F, Holsboer F, Rupprecht R. Allopregnanolone affects sleep in a benzodiazepine-like fashion. Journal of Pharmacology & Experimental Therapeutics 1997; 282(3):1213-1218. Montplaisir J, Lorrain J, Denesle R, Petit D. Sleep in menopause: differential effects of two forms of hormone replacement therapy. Menopause 2001;10-16. Steiger A, Trachsel L, Guldner J, Hemmeter U, Rothe B, Rupprecht R, Vedder H, Holsboer F. Neurosteroid pregnenolone induces sleep-EEG changes in man compatible with inverse agonistic GABAA-receptor modulation. Brain Research 1993; 615:267-274.